CLINICAL TRIAL: NCT01600716
Title: Safety and Efficacy Study of OnabotulinumtoxinA for the Treatment of Urinary Incontinence Due to Neurogenic Detrusor Overactivity (NDO) in Non-Catheterizing Patients With Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-117
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Urinary Incontinence; Multiple Sclerosis; Neurogenic Bladder
MeSH Terms: conditions — Urinary Incontinence; Multiple Sclerosis; Urinary Bladder, Neurogenic | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OnabotulinumtoxinA (Experimental): OnabotulinumtoxinA 100 U is administered into the detrusor at Day 1. After a minimum of 12 weeks, patients could request/qualify for a second onabotulinumtoxinA 100 U injection.
  Interventions: Biological: OnabotulinumtoxinA
- Placebo (Normal Saline) (Other): Placebo (normal saline) is administered into the detrusor at Day 1. After a minimum of 12 weeks, patients could request/qualify for an onabotulinumtoxinA injection.
  Interventions: Biological: OnabotulinumtoxinA; Drug: Placebo (Normal Saline)

INTERVENTIONS:
Biological: OnabotulinumtoxinA — OnabotulinumtoxinA 100 U is administered into the detrusor at Day 1 in the onabotulinumtoxinA 100 U arm. After a minimum of 12 weeks, patients in both the onabotulinumtoxinA 100 U arm and the placebo arm could request/qualify for an onabotulinumtoxinA injection.
  Other Names: BOTOX®; botulinum toxin Type A
Drug: Placebo (Normal Saline) — Placebo (normal saline) is administered into the detrusor at Day 1.
  Arms: Placebo (Normal Saline)

SUMMARY:
This study will evaluate the safety and efficacy of OnabotulinumtoxinA (BOTOX®) for the treatment of urinary incontinence due to NDO in non-catheterizing patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 episodes of urinary incontinence over a 3-day period
* History of Multiple Sclerosis (MS)
* Urinary incontinence not adequately controlled by anticholinergic medication

Exclusion Criteria:

* Current use of intermittent catheter or indwelling catheter to manage urinary incontinence
* Previous or current botulinum toxin therapy of any serotype for any urological condition
* Previous or current botulinum toxin therapy of any serotype for any non-urological condition within the last 12 weeks
* Diagnosis of myasthenia gravis, Eaton-Lambert Syndrome, or Amyotrophic Lateral Sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2012-06-13 (Actual); Primary Completion 2014-04-04 (Actual); Study Completion 2015-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (10):
- Mountlake Terrace, Washington, United States
- Liège, Belgium
- Canada (2):
  - Victoria, British Columbia
  - Kitchener, Ontario
- Olomouc, Czechia
- France (2):
  - Garches
  - Marseille
- Warsaw, Poland
- Porto, Portugal
- Saint Petersburg, Russia

REFERENCES:
- [Background] Tullman M, Chartier-Kastler E, Kohan A, Keppenne V, Brucker BM, Egerdie B, Mandle M, Nicandro JP, Jenkins B, Denys P. Low-dose onabotulinumtoxinA improves urinary symptoms in noncatheterizing patients with MS. Neurology. 2018 Aug 14;91(7):e657-e665. doi: 10.1212/WNL.0000000000005991. Epub 2018 Jul 20. PMID 30030330

RESULTS

PARTICIPANT FLOW:
Groups:
- OnabotulinumtoxinA: OnabotulinumtoxinA 100 U is administered into the detrusor at Day 1. After a minimum of 12 weeks, patients could request/qualify for a second onabotulinumtoxinA injection.
Period: Overall Study
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Started | 66 | 78
Completed | 59 | 71
Not Completed | 7 | 7
Not completed — Other Reasons | 3 | 1
Not completed — Personal Reasons | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Lack of Efficacy | 2 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 66 | 78 | 144
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 62 | 71 | 133
  ≥65 years | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 70 | 127
  Male | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Average Frequency of Urinary Incontinence Episodes
Description: Incontinence is defined as involuntary loss of urine as recorded in a patient bladder diary. The number of episodes of urinary incontinence is recorded over a 3-day period the week of the study visit. A negative number change from baseline indicates a reduction in incontinence episodes (improvement) and a positive number change indicates an increase in incontinence episodes (worsening).
Time Frame: Baseline, Week 6
Population: Intent-to-Treat Population: all randomized patients
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 66 | 78
Episodes
  Baseline | 4.18 (3.167) | 4.32 (2.422)
  Change from Baseline at Week 6 | -3.34 (2.881) | -1.10 (2.083)

2. Secondary Outcome: Change From Baseline in Maximum Cystometric Capacity (MCC)
Description: MCC represents the maximum volume of urine the bladder holds. A positive number change from baseline represents an improvement (increase) in the maximum volume of urine the bladder holds and a negative number change from baseline represents a worsening (decrease) in the maximum volume of urine the bladder holds.
Time Frame: Baseline, Week 6
Population: Intent-to-Treat Population: all randomized patients with data at the time points
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 65 | 78
Milliliters (mL)
  Baseline | 246.4 (138.49) | 245.7 (133.90)
  Change from Baseline at Week 6 (N=62,72) | 127.2 (139.25) | -1.8 (93.23)

3. Secondary Outcome: Change From Baseline in Maximum Detrusor Pressure During the First Involuntary Detrusor Contraction (IDC)
Description: Maximum detrusor pressure represents the maximum pressure (peak amplitude) in the bladder during the first involuntary contraction of the bladder muscle. A negative number change from baseline indicates an improvement in pressure and a positive number change from baseline indicates a worsening in pressure.
Time Frame: Baseline, Week 6
Population: Intent-to-Treat Population: all randomized patients with data at the time points
Measure: Mean (Standard Deviation); unit: Centimeters of Water (cm H2O)
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 57 | 69
Centimeters of Water (cm H2O)
  Baseline | 35.9 (34.90) | 36.1 (37.21)
  Change from Baseline at Week 6 (N=25,51) | -19.6 (37.61) | 3.7 (33.24)

4. Secondary Outcome: Change From Baseline in Incontinence Quality of Life Instrument (I-QOL) Total Summary Score
Description: The I-QOL is a validated, disease-specific quality of life (QOL) questionnaire containing 22 questions designed to measure impact of urinary incontinence on patients' lives. Each question is answered on a 5-point scale (1 = worst QOL, and 5 = best QOL). The scores are totaled over the 22 questions and normalized to a score of 0-100 (0=worst QOL and 100=best QOL). A positive change from baseline represents an improvement and a negative change from baseline represents a worsening.
Time Frame: Baseline, Week 6
Population: Intent-to-Treat Population: all randomized patients with data at the time points
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 58 | 74
Scores on a Scale
  Baseline | 32.43 (16.337) | 34.24 (21.163)
  Change from Baseline at Week 6 (N=55,68) | 40.39 (26.499) | 9.92 (15.863)

5. Other Pre Specified Outcome: Duration of Treatment Effect Through Week 52
Description: The duration of treatment effect is the time to patient request for retreatment.
Time Frame: Up to 52 Weeks
Population: Intent-to-Treat Population: all randomized patients
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 66 | 78
Weeks | 51.7 [36.9 to NA] — The upper confidence limit was not estimable since too few patients had requested retreatment prior to the end of the study. | 12.6 [12.3 to 13.0]

ADVERSE EVENTS:
Description: Adverse events and serious adverse events are analyzed by treatment cycle (cycle 1 and cycle 2).
Groups:
- OnabotulinumtoxinA Treatment Cycle 1: OnabotulinumtoxinA 100 U is administered into the detrusor at Day 1. Median duration of exposure is 50.7 weeks.
- Placebo (Normal Saline): Placebo (normal saline) is administered into the detrusor at Day 1. Median duration of exposure is 15.2 weeks.
- OnabotulinumtoxinA/OnabotulinumtoxinA Treatment Cycle 2: OnabotulinumtoxinA 100 U is administered into the detrusor at Day 1. After a minimum of 12 weeks, a second onabotulinumtoxinA injection is given. Median duration of exposure is 12.5 weeks.
- Placebo (Normal Saline)/OnabotulinumtoxinA: Placebo (normal saline) is administered into the detrusor at Day 1. After a minimum of 12 weeks, an onabotulinumtoxinA injection is given. Median duration of exposure is 12.2 weeks.
Arm/Group | OnabotulinumtoxinA Treatment Cycle 1 | Placebo (Normal Saline) | OnabotulinumtoxinA/OnabotulinumtoxinA Treatment Cycle 2 | Placebo (Normal Saline)/OnabotulinumtoxinA
Serious Adverse Events (participants affected / at risk) | 7/66 | 3/78 | 0/30 | 2/67
Other Adverse Events (participants affected / at risk) | 50/66 | 44/78 | 21/30 | 38/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA Treatment Cycle 1 (N=66) | Placebo (Normal Saline) (N=78) | OnabotulinumtoxinA/OnabotulinumtoxinA Treatment Cycle 2 (N=30) | Placebo (Normal Saline)/OnabotulinumtoxinA (N=67)
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 0 | 0 | 0
Infectious Colitis (Infections and infestations) | 0 | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 — Onset date was 135 days after administration of onabotulinumtoxinA
Multiple Sclerosis Relapse (Nervous system disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA Treatment Cycle 1 (N=66) | Placebo (Normal Saline) (N=78) | OnabotulinumtoxinA/OnabotulinumtoxinA Treatment Cycle 2 (N=30) | Placebo (Normal Saline)/OnabotulinumtoxinA (N=67)
Urinary tract infection (Infections and infestations) | 26 | 9 | 9 | 17
Urinary Retention (Renal and urinary disorders) | 11 | 3 | 6 | 9
Residual Urine Volume (Investigations) | 11 | 2 | 1 | 5
Bacteriuria (Infections and infestations) | 12 | 6 | 3 | 6
Leukocyturia (Renal and urinary disorders) | 4 | 6 | 1 | 2
Dysuria (Renal and urinary disorders) | 6 | 1 | 3 | 1
Haematuria (Renal and urinary disorders) | 3 | 6 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 0 | 0
Renal Cyst (Renal and urinary disorders) | 3 | 3 | 3 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 0
Micturition Urgency (Renal and urinary disorders) | 2 | 0 | 2 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 0 | 2 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 2 | 0
Urine Abnormality (Renal and urinary disorders) | 1 | 0 | 2 | 0
Urine Odour Abnormal (Renal and urinary disorders) | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.